CLINICAL TRIAL: NCT02325648
Title: The Intraoperative Physiologic Changes of Patients Under Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Cytoreductive Surgery; Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0854
Record Dates: First submitted 2014-12-14; First posted 2014-12-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Peritoneal Surface Malignancies
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIPEC cytoreductive surgery
  Interventions: Drug: HIPEC cytoreductive surgery

INTERVENTIONS:
Drug: HIPEC cytoreductive surgery — At least 30 minutes prior to the prospective conclusion of the surgery, 1 μg/kg of fentanyl is administered for postoperative analgesia and 0.075mg of palonosetron is IV-infused for the prevention of nausea and vomiting. Desflurane and remifentanil administration is ceased after the surgery is concluded, muscle relaxation is evaluated by train of four (TOP) monitoring using a nerve stimulator, and the neuromuscular blockade is reversed with 0.2 mg of glycopyrrolate and 1 mg of neostigmine. When the patient recovers consciousness and begins spontaneous respiration, extubation is performed and the patient is transferred to the ICU with monitoring of their vital signs.

SUMMARY:
The most popular surgical treatment of peritoneal cancer is the type known as hyperthermic intraperitoneal chemoperfusion (HIPEC), a type of cytoreductive surgery for which a significantly high survival rate has been demonstrated by several studies. It is widely known that HIPEC entails severe physiological changes and precautions during anesthesia. However, very few studies have systematically outlined and organized these changes for each system, and most existing studies only report retrospective data or are limited to gynecological surgeries. Therefore, the present researchers planned a prospective observational study to determine the physiological changes that occur in patients during HIPEC cytoreductive surgeries performed in the colon and rectal surgery department of the investigators hospital. The investigators planned to monitor the patients' body temperature, metabolism, cardiovascular and respiratory changes during HIPEC cytoreductive surgery and analyze the anesthetic methods applied to identify the optimal anesthetic management strategy for HIPEC cytoreductive surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 20 years of age or older who will undergo HIPEC cytoreductive surgery at the colon and rectal surgery department of our hospital

Exclusion Criteria:

* Cases in which there is a sudden change of surgery plans, or those in which consent forms are retracted.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who undergoing HIPEC cytoreductive surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Vital sign | from 30 minutes to 90 minutes after HIPEC
Body temperature | from 30 minutes to 90 minutes after HIPEC
serum glucose | from 30 minutes to 90 minutes after HIPEC
pulmonary vascular permeability index | from 30 minutes to 90 minutes after HIPEC

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea, South Korea

REFERENCES:
- [Derived] Kim MH, Yoo YC, Bai SJ, Lee KY, Kim N, Lee KY. Physiologic and hemodynamic changes in patients undergoing open abdominal cytoreductive surgery with hyperthermic intraperitoneal chemotherapy. J Int Med Res. 2021 Jan;49(1):300060520983263. doi: 10.1177/0300060520983263. PMID 33445991